CLINICAL TRIAL: NCT06028334
Title: GetUp&Go: A Randomized Controlled Trial of a Theory-Based Intervention to Enhance Physical Activity in Chronic, Moderate-Severe Traumatic Brain Injury
Brief Title: GetUp&Go: A Randomized Controlled Trial of an Intervention to Enhance Physical Activity After TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Rabinowitz, Institute Scientist, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iRISID-2023-1533
Record Dates: First submitted 2023-03-02; First posted 2023-09-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: physical activity; mobile health
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a waitlist controlled randomized trial. All participants will receive the GetUp&Go treatment program. Participants will be randomly assigned with a 50% chance of either receiving immediate treatment (IT) with the 10-week program, or going on a 10-week waitlist, after which they will start the GetUp&Go program.
Who Masked: Outcomes Assessor
Masking Description: This project will use masked outcome assessment, with special precautions taken to prevent inadvertent unmasking. These include a "script" reminding participants not to discuss any of their experiences in the trial. Any instances of inadvertent unmasking will be recorded for later analysis of their influence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (Experimental): The 10-week GetUp&Go intervention will be delivered entirely remotely, with 2 weekly sessions with a therapist delivered over videoconference (Zoom for Healthcare) followed by 3 sessions in weeks 3, 5, and 8, over Zoom or phone according to participant preference.
  The overall goal of the intervention is to develop and support a personalized plan to increase physical activity and decrease sedentary behavior, in concert with the unique capabilities, opportunities, and motivational factors of each participant. In session 2 and thereafter, RehaBot will be supplied to participants to deliver therapeutic ingredients to supplement those provided by the therapist.
  Interventions: Behavioral: GetUp&Go
- Waitlist (Placebo Comparator): A 10-week waitlist with baseline and outcome assessment, followed by receipt of the full GetUp&Go program.
  Interventions: Behavioral: GetUp&Go with 10-Week Delay

INTERVENTIONS:
Behavioral: GetUp&Go — A behavioral treatment combining personalized activity planning and a mobile health application for supporting adherence to activity plans.
  Arms: Immediate Treatment
Behavioral: GetUp&Go with 10-Week Delay — No assigned treatment during the waitlist phase. Participants in the WL group will be offered the GetUp&Go intervention, which combines personalized activity planning and a mobile health application, after collection of the primary outcome measure.
  Arms: Waitlist

SUMMARY:
The goal of this clinical trial is to evaluate GetUp&Go, a program for promoting increased physical activity in individuals at least 6 months post moderate-to-severe traumatic brain injury. GetUp&Go is a remotely delivered 10-week program that includes one-on-one sessions with a therapist and a mobile health application (RehaBot).

The main question is whether participants in the 10-week GetUp&Go program increase their physical activity, and exhibit associated benefits in mental and physical health, relative to those who are put on a waitlist.

* Question 1: Do participants who receive immediate treatment with GetUp&Go show more increased physical activity, measured by accelerometer activity counts per day, and improve more on secondary outcomes, such as self-reported physical activity, emotional function, fatigue, sleep, pain, and health-related quality of life, compared to their baseline, relative to those who are put on a waitlist?
* Question 2: Do participants who have continued access to the mobile health component of the intervention, RehaBot, show better maintenance of physical activity gains compared to those who no longer have access to RehaBot?
* Question 3: Are individual participant characteristics associated with participants' response to the treatment program?

DETAILED DESCRIPTION:
The investigators will conduct a Randomized Controlled Trial (RCT) of a novel, remotely delivered physical activity (PA) promotion program, called GetUp&Go-a name selected by focus group participants with moderate-to-severe traumatic brain injury (msTBI). It will be theoretically based, use objective measurement of PA as a primary outcome, and incorporate varied types and amounts of home- and neighborhood-based PA and ways to reduce sedentary behavior, according to participant preferences. Moreover, using a 2-phase design as described below, the investigators will test a method for enhancing longer-term gains in PA using mobile technology, in addition to gains acquired during the first phase of intervention.

Trial design. Participants will undergo baseline testing (T1) and will then be randomized 1:1 to either immediate treatment in GetUp&Go (IT) or waitlist (WL) for 10 weeks. After testing for the primary outcome (T2), the waitlist group will receive GetUp&Go for 10 weeks followed by a T2b evaluation for that group. This phase is called the "A phase", for Acquisition.

Following completion of the GetUp&Go intervention, all participants-regardless of initial group allocation-will be randomized 1:1 to one of two conditions for an additional 10 weeks, the "Follow-Through" (FT) phase. Half of participants will be randomized to the RehaBot condition (RB), which provides continued use of the chatbot to support individualized PA plans, but with no further therapist contact. Participants in the No RehaBot (No RB) condition will not have access to the chatbot. The final evaluation, T3, will occur after the 10-week Follow-Through phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* TBI (open or closed), sustained at least 6 months prior to enrollment, of at least complicated-mild/moderate severity as evidenced by loss or alteration of consciousness ≥ 30 minutes; and/or post-traumatic amnesia (PTA) ≥ 24 hours, not due to intoxication/sedation and documented prospectively from the injury; and/or positive neuroimaging findings consistent with TBI
* Fully weight bearing on lower limbs and able to walk indoors and outdoors without the assistance of another person
* Cognitively able to participate in treatment as judged by ability to travel independently within the community
* Able to communicate adequately in English for participation in the treatment protocols
* Informed consent given by participant

Exclusion Criteria:

* Contraindications to increasing PA as judged by study physician, using an exam based on published screening tools
* Medical or psychiatric instability, including current psychosis or severe uncontrolled substance misuse, as assessed using items from the SCID/MINI/ASSIST, or suicidal ideation with intent or plan, as assessed by the Columbia-Suicide Severity Rating Scale, screening version
* Significant physical or intellectual disability predating the TBI
* Neurodegenerative disorder, e.g., Parkinson's disease
* Insufficiently inactive, i.e., reporting > 23 weekly moderate/vigorous activity units on the Godin Leisure-Time Exercise Questionnaire
* Planned surgery or other hospitalization during the succeeding 9 months
* Physical or sensory disability (e.g., blindness; severe bimanual incoordination) that prevents use of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Average activity counts/minute | Baseline
  Actigraphy derived average activity counts/minute from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Average activity counts/minute | 10 weeks after initial randomization
  Actigraphy derived average activity counts/minute from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Average activity counts/minute | 10 weeks after completing GetUp&Go intervention
  Actigraphy derived average activity counts/minute from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period

SECONDARY OUTCOMES:
Percent (%) time sedentary | Baseline
  Actigraphy derived percent time sedentary from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Percent (%) time sedentary | 10 weeks after initial randomization
  Actigraphy derived percent time sedentary from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Percent (%) time sedentary | 10 weeks after completing GetUp&Go intervention
  Actigraphy derived percent time sedentary from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Percent (%) time engaged in moderate-vigorous physical activity (MVPA) | Baseline
  Actigraphy derived percent time engaged in MVPA from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Percent (%) time engaged in moderate-vigorous physical activity (MVPA) | 10 weeks after initial randomization
  Actigraphy derived percent time engaged in MVPA from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Percent (%) time engaged in moderate-vigorous physical activity (MVPA) | 10 weeks after completing GetUp&Go intervention
  Actigraphy derived percent time engaged in MVPA from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Average daily step count | Baseline
  Actigraphy derived average daily step count from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Average daily step count | 10 weeks after initial randomization
  Actigraphy derived average daily step count from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Average daily step count | 10 weeks after completing GetUp&Go intervention
  Actigraphy derived average daily step count from wrist-worn Actigraph GT3XP averaged over 4 consecutive-wear days over a 7-day period
Self-reported PA | Baseline
  Physical Activity Scale for Individuals with Physical Disabilities (Scale: 0-100, where higher scores indicate a greater level of activity)
Self-reported PA | 10 weeks after initial randomization
  Physical Activity Scale for Individuals with Physical Disabilities (Scale: 0-100, where higher scores indicate a greater level of activity)
Self-reported PA | 10 weeks after completing GetUp&Go intervention
  Physical Activity Scale for Individuals with Physical Disabilities (Scale: 0-100, where higher scores indicate a greater level of activity)
Emotional function | Baseline
  Brief Symptom Inventory-18 (Scale: 0-72, where higher scores indicate the presence of more psychiatric symptoms)
Emotional function | 10 weeks after initial randomization
  Brief Symptom Inventory-18 (Scale: 0-72, where higher scores indicate the presence of more psychiatric symptoms)
Emotional function | 10 weeks after completing GetUp&Go intervention
  Brief Symptom Inventory-18 (Scale: 0-72, where higher scores indicate the presence of more psychiatric symptoms)
Fatigue | Baseline
  Fatigue Severity Scale Short Form (Scale: 9-63, where higher scores indicate greater fatigue)
Fatigue | 10 weeks after initial randomization
  Fatigue Severity Scale Short Form (Scale: 9-63, where higher scores indicate greater fatigue)
Fatigue | 10 weeks after completing GetUp&Go intervention
  Fatigue Severity Scale Short Form (Scale: 9-63, where higher scores indicate greater fatigue)
Sleep Quality | Baseline
  Pittsburgh Sleep Quality Index (Scale: 0-21, where higher scores indicate poorer sleep quality)
Sleep Quality | 10 weeks after initial randomization
  Pittsburgh Sleep Quality Index (Scale: 0-21, where higher scores indicate poorer sleep quality)
Sleep Quality | 10 weeks after completing GetUp&Go intervention
  Pittsburgh Sleep Quality Index (Scale: 0-21, where higher scores indicate poorer sleep quality)
Subjective pain | Baseline
  Brief Pain Interference Scale (Scale: 6-30, where higher scores indicate greater pain interference)
Subjective pain | 10 weeks after initial randomization
  Brief Pain Interference Scale (Scale: 6-30, where higher scores indicate greater pain interference)
Subjective pain | 10 weeks after completing GetUp&Go intervention
  Brief Pain Interference Scale (Scale: 6-30, where higher scores indicate greater pain interference)
Health-related Quality of Life | Baseline
  Quality of Life after Brain Injury Scale (Scale: 0-100, where higher scores indicate better quality of life)
Health-related Quality of Life | 10 weeks after initial randomization
  Quality of Life after Brain Injury Scale (Scale: 0-100, where higher scores indicate better quality of life)
Health-related Quality of Life | 10 weeks after completing GetUp&Go intervention
  Quality of Life after Brain Injury Scale (Scale: 0-100, where higher scores indicate better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rabinowitz, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected for this trial will be submitted the Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system.
  The data submitted to FITBIR will be fully de-identified and contain the Global Unique Identifier (GUID). The investigators will assign GUIDs to cases using the methodology recommended by FITBIR. If it is not possible to assign a GUID to cases, a Pseudo-GUID will be assigned. All variables will be converted to the TBI Common Data Elements (CDEs), to the extent possible; otherwise variables that do not map to the TBI CDEs will be submitted as Unique Data Elements (UDEs).
Supporting Information: Study Protocol
Time Frame: All data from this trial will be submitted to FITBIR within one year of the completion of the award, per the FITBIR submission schedule for clinical trials.
Access Criteria: Projects must be specified for research purposes only (not commercial) with the intention to enhance knowledge for the benefit of human health.
  Individuals requesting access must have a medical or scientific degree or position relevant for the request.
  Individuals must be affiliated with a research, industry, or non-profit institution/business/organization.
  All data access requests must be signed by an individual legally authorized to sign on behalf of the institution/business/organization.
URL: https://fitbir.nih.gov/